CLINICAL TRIAL: NCT05326568
Title: The Effect of Sesame Oil on the Prevention of Phlebitis in Patients Undergoing Cardiac Surgery
Brief Title: Effect of Sesame Oil in Preventing Phlebitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Muaz Gulsen, Academic Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CukurovaUnıversıty-Mgulsen-01
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Phlebitis After Infusion
Keywords: aromatherapy; amiodarone infusion; phlebitis; cardiac surgery; Sesame oil
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: After the research report is written, a third person will assign an intervention and control group to the letters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Sesame oil was applied by the researcher to the patients assigned to the intervention group. Sesame oil was applied to the 10 cm circumference of the cannula, in the form of 10 drops and 10 minutes.
  Interventions: Other: Complementary treatment practice
- Control (No Intervention): No treatment was applied to the patients assigned to the control group and only standard care was applied.

INTERVENTIONS:
Other: Complementary treatment practice — Applying sesame oil to the patients assigned to the intervention group by applying 10 drops to the 10 cm circumference of the cannula for 10 minutes
  Arms: Experimental

SUMMARY:
Background: To determine the effect of sesame oil in preventing phlebitis that may occur during intravenous therapy in patients undergoing cardiac surgery.

Material and Method: A randomized controlled interventional study will be conducted with patients treated in the coronary intensive care unit of a university hospital. The population of the study will be the patients hospitalized in the intensive care unit after cardiac surgery and administered parenteral amiodarone infusion. The power analysis was carried out by taking the study by. The sample size was determined as 44 patients. Personal Information Form and Visual Infusion Phlebitis Scale will be used to collect data. Sesame oil will be applied to the patients in the intervention group as 10 drops, 10 cm around the cannula, for 10 minutes. This administration will be repeated every eight hours during the 24-hour amiodarone infusion. No application will be made by the researcher to the patients in the control group. At the end of each 24 hours, patients in both groups will be evaluated by the investigator on the Visual Infusion Phlebitis Scale. Descriptive statistics, chi square, independent t test and Fisher's exact test will be used to evaluate the data.

DETAILED DESCRIPTION:
No application was made to the patients assigned to the control group. Sesame oil was applied by the researcher to the patients assigned to the intervention group. Sesame oil was applied to the 10 cm circumference of the cannula by applying 10 drops and 10 minutes. This application was repeated every eight hours during the 24-hour amiodarone infusion. The area where the intravenous line is located is covered with a standard transparent dressing (Tegaderm) so that it can be observed. Patients in the intervention and control groups were evaluated for phlebitis at the end of every 24 hours (1st day, 2nd day, 3rd day) according to the VIP scale. The highest of the phlebitis stages obtained as a result of the evaluation was accepted as the final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone cardiac surgery,
* were over 18 years old,
* were conscious, could communicate,
* were not allergic to sesame,
* were administered prophylactic rhythm regulator
* amiodarone as a treatment were included in the study.

Exclusion Criteria:

* who was with cancer,
* who was with diabetes mellitus,
* who was with hypertension
* who was with peripheral vascular disease
* Patients who had myocardial infarction during the procedure,
* Received immunosuppressive therapy,
* underwent resuscitation and could not use an intravenous catheter for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Visual Infusion Phlebitis Scale | Change from 1st day to 2nd day, and 3rd day after the implementation
  The scale monitors the potential risks of the catheter when administering peripheral venous therapy and rates the developmental stages of phlebitis. Scores range from 0-4. A score of zero indicates that there are no signs of phlebitis, and a score of four indicates that the phlebitis is in the last stage.

CONTACTS AND LOCATIONS:
Overall Officials: Sevban ARSLAN, PhD, Study Director — Cukurova University
Locations (1):
- Muaz GÜLŞEN, Adana, Turkey (Türkiye)